CLINICAL TRIAL: NCT06591143
Title: Evaluation Of Periodontal Health After Treatment With Hall Technique Compared to Atraumatic Restorative Treatment in The Management of Carious Primary Molars: A Randomized Clinical Trial
Brief Title: Evaluation Of Periodontal Health After Treatment With Hall Technique Versus Atraumatic Restorative Treatment in The Management of Carious Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Medhat, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT Vs ART
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Decayed Primary Molars
Keywords: Decayed primary molars ART Hall technique

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART (Experimental): Atraumatic restorative treatment
  Interventions: Procedure: ART
- Hall technique (Experimental): Stainless steel crown placement without tooth preparation
  Interventions: Procedure: Hall technique

INTERVENTIONS:
Procedure: ART — Caries excavation with hand instruments only and restoration with glass ionomer filling
  Arms: ART
Procedure: Hall technique — Stainless steel crown placement without tooth preparation
  Arms: Hall technique

SUMMARY:
This trial seeks to evaluate the periodontal health of two modalities Hall Technique (by placing a stainless steel crown without caries removal, local anaesthesia won't be needed) & ART (by removing caries by sharp excavator and restoring the tooth with glass ionomer, local anaesthesia won't be needed either) to achieve better treatment for caries with pain-free procedures in developing countries that have high caries index and low income.

ELIGIBILITY:
Inclusion Criteria:

* Age: From 4 to 6 years.
* Caries in primary molars within enamel/dentin with vital pulp.
* Healthy children.
* Cooperative children.

Exclusion Criteria:

* Presence of signs and symptoms of necrosis.
* Root caries.
* History of Spontaneous pain.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal health | initial, 3 months, 6 months, 12 months
  While determining the plaque, the 4 surfaces of the teeth included in the study (mesial, distal, vestibule, lingual) using plaque index (0: no plaque, 2: thick visible plaque easily detected)

SECONDARY OUTCOMES:
Gingival index | Initial, 3 months, 6 months, 12 months
  While determining the plaque, the 4 surfaces of the teeth included in the study (mesial, distal, vestibule, lingual) (0= no swelling, 2= Moderate to severe gingival swelling, bleeding after air drying)
Postoperative pain and discomfort | Immediately postoperative
  Immediately after the treatment, any pain and discomfort experienced by the child will be recorded using the Face Pain Scale - revised (FPS-R) (0= no pain, 10=worst)
Child behaviour | Intraoperative
  Venham Anxiety Rating Scale (0= total cooperation, best possible working conditions, no crying or physical protest, 5= general protest, no cooperation, physical restraint is required)
Child anxiety | Intraoperative
  Venham Anxiety Rating Scale (0= relaxed, smiling, willing, and able to converse, 5= loud crying unable to listen to verbal communication)
Canine overbite | Initial, 3 months, 6 months, 12 months
  The canine overbite will be calculated before the preparation by measuring the distance between the incisal points of the maxillary canine on the same side of the mouth to the gingival zenith of the mandibular canine using a Boley Gauge

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR